CLINICAL TRIAL: NCT06082427
Title: Virtual Reality Hypnosis Prior to Radiofrequency Thermocoagulation for Patients With Chronic Pain: A Prospective Quasi-Randomized Controlled Trial
Brief Title: Impact of Virtual Reality Hypnosis Before an Invasive Medical Procedure for Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: /344
Record Dates: First submitted 2023-09-12; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain
Keywords: Virtual reality hypnosis; Radiofrequency thermocoagulation; Chronic pain; Anxiety; Complementary approach
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRH (Experimental): VRH was delivered through a 3D virtual reality headpiece equipped with a head-tracking system called " IPNEO " and designed by the society Cayceo (Montpellier, France, https://cayceo.fr/). The device display an enchanted environment movie based on hypnosis induction and suggestions (relaxation, comfort, and safety).
  Interventions: Device: Virtual reality hypnosis
- Control (No Intervention): Usual care

INTERVENTIONS:
Device: Virtual reality hypnosis — VRH was delivered through a 3D virtual reality headpiece equipped with a head-tracking system based on hypnosis induction and suggestions (relaxation, comfort, and safety). The complete intervention lasted 17 minutes.
  Arms: VRH

SUMMARY:
Management of chronic pain involves an array of tools, such as radiofrequency thermocoagulation (Rf-Tc). Like many other invasive procedures, Rf-Tc can generate an increase in pain perception and anxiety levels. Virtual reality hypnosis (VRH) is a promising tool in managing anxiety and pain. Nevertheless, its effectiveness has not been investigated in patients with chronic pain goig througha Rf-Tc procedure. The goal of this study is to evaluate the effectiveness of VRH on self-assessed anxiety in patients with chronic pain having to undergo an act of Tf-Rc. Patients were randomly assigned into two groups: VRH or Control (usual care). Assessment were carried-out at 4 periods of time: T0 (the week before the Rf-Tc); T1 (pre-intervention the day of the Rf-Tc); T2 (post-intervention the day of the Rf-Tc); and T3 (post-Rf-Tc). Medical and socio-demographic data, immersive tendencies pain, anxiety, and satisfaction were assessed at each time points.

ELIGIBILITY:
Inclusion Criteria:

* suffering from chronic pain
* >18 years old
* French speaking
* no claustrophobia
* no head or face wounds
* sufficient auditory and visual acuity for an effective use of the VRH technique

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Anxiety | One week before the Radiofrquency; on the day of the radiofrequency before the VRH/Ctr; right after the VRH/Ctr, and after the radiofrequency
  Assessed with a numerical rating scale (0= no anxiety; 10= worst anxiety).

SECONDARY OUTCOMES:
Anxiety trait | One week before the Radiofrquency
  Assessed with the State-Trait Anxiety Inventory. This questionnaire includes 20 items assessing trait anxiety The scores can vary from 20 to 80. The higher the score, the more the individual is said to be anxious
Pain intensity | One week before the Radiofrquency; on the day of the radiofrequency before the VRH/Ctr; right after the VRH/Ctr, and after the radiofrequency
  Assessed with a numerical rating scale (0= no pain; 10= worst pain immaginable).
Immersive tendencies | On the day of the radiofrequency before the VRH/Ctr
  Immersive tendencies questionnaire contains 18 items rated on a scale of 1 (never) to 7 (often). It contains 4 sub-scales : "Focus" is the tendency to stay focused on ongoing activities; "Involvement" is the tendency to become involved in activities ; "Emotion" is the tendency to be emotionally involved by the environment; "Game" is the tendency to play video games. A total score is also available, and it varies from 18 to 126. The higher the score, the higher the tendency for immersion in the virtual environment.
Sens of presence | Right after the VRH/Ctr
  The 12-item Presence Questionnaire is a self-made questionnait that assesses patients' feelings during the experience in the immersive environment. All items are rated from 1 to 7 The higher the scores, the more impressions experienced by the participants are perceived as real.
Satisfaction | After the radiofrequency, Average 1 hour
  Assessed with a numerical rating scale (0= total dissatisfaction, 10= total satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No